CLINICAL TRIAL: NCT01558284
Title: Clinical Study on the Effect of Neu-P11 on Symptoms in Patients With Diarrhea- Irritable Bowel Syndrome (D-IBS)
Brief Title: The Effect of Neu-P11 on Symptoms in Patients With D-IBS
Acronym: Neu-P11
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Martin Storr, Prof Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: STO-010; 2011-002657-60 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-20 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Diarrhea- Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Neu-P11; Melatonin; D-IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — N-(2-(5-methoxy-indol-3-yl)-ethyl)-4-oxo-4H-pyran-2-carboxamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Neu-P11 — Neu-P11 is a new Melatonin receptor-, Serotonin 5-HT- 1A and 5-HT- 1D - agonist and a serotonin 5-HT- 2B - antagonist
  Other Names: there are no other names
Drug: Placebo — Placebo
  Other Names: there are no other names

SUMMARY:
Placebo controlled double-blind study with 40 patients who have an diarrhea-predominant IBS, 20 get Neu-P11, 20 get a placebo. Neu-P11 is a, Melatonin receptor-, Serotonin 5-HT- 1A and 5-HT- 1D - agonist and a serotonin 5-HT- 2B - antagonist.

DETAILED DESCRIPTION:
This study aims to test a possible beneficial effect of NEU-P11 in patients with IBS.

The effect on symptoms will be rated by symptom scores. The primary endpoint will be the symptomatic benefit reported by the patient answering the simple question: Did your symptoms improve compared to prior to the clinical trial.

Additional secondary endpoints will capture sleep quality, changes in stool texture and individual symptom scores employing standardized symptom scores.

The study design is a 4 week, randomised, placebo-controlled, double blind study where 40 patients receive either placebo (20) or NEU-P11 (20). In the mid of the four week time of the Study the dose can be doubled of the patient does not recognize any relief of the D-IBS.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18-80 years old
2. Male or female

   Women of childbearing potential must have a negative pregnancy test at the screening visit, on Day 1 of each treatment period, and use a reliable method of contraception during the entire study duration and for at least 3 months after study drug intake. Reliable methods of contraception are:
   * oral contraception
   * Double barrier type devices (e.g., male or female condom, diaphragm, contraceptive sponge) only in combination with a spermicide.
   * Intra-uterine devices in combination with a spermicide. Abstention, rhythm method, and contraception by the partner alone are not acceptable methods of contraception. Women not of childbearing potential are defined as postmenopausal (i.e., amenorrhea for at least 1 year), or surgically or naturally sterile.
3. Subject has IBS confirmed by the Rome III diagnostic criteria

Exclusion Criteria:

1. Subject has current evidence of duodenal ulcer, gastric ulcer, diverticulitis, or infectious gastroenteritis.
2. Subject has a history of inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis, celiac disease), GI malignancy, GI obstruction, gastroparesis, carcinoid syndrome, pancreatitis, amyloidosis or ileus
3. Subject is a candidate for GI surgery or has a history of GI surgery except appendectomy and cholecystectomy.
4. Subject has psychiatric disorders which are not controlled (based on the investigator medical judgment); subject with psychosis are excluded regardless of current therapy.
5. Subject has current or recent history (within 12 months of signing on informed consent) of drug or alcohol abuse.
6. Subject is pregnant or lactating
7. Subject has history of human immunodeficiency virus (HIV) or hepatitis (B or C)
8. Subject has any condition or circumstance that could cause noncompliance with treatments or visits
9. Subject has active malignancy within the last 5 years.
10. Subject taking antipsychotic drugs, antispasmodics, antidiarrheals (e.g. loperamide, lubiprostone and bismuth subsalicylate), narcotics, prokinetic drugs, drugs indicated for IBS (e.g Alosetron), or warfarin.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diarrhea-praedominant Irritated Bowel Syndroms
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The relief of symptoms of the D-IBS by the study medication. | after each week for the time of study
  Only one question at the end of each visit and of each telephone call

CONTACTS AND LOCATIONS:
Overall Officials: Martin Storr, Prof Dr., Principal Investigator — Medizinische Klinik 2 LMU Muenchen
Locations (1):
- Klinikum Grosshadern Medizinische Klinik 2, Munich, Bavaria, Germany

REFERENCES:
- [Background] Storr M. [Therapy of gastroesophageal reflux disease (GERD)]. Med Monatsschr Pharm. 2011 Dec;34(12):446-54; quiz 455-6. German. PMID 22233024
- See also: Sponsor of the Trial — http://www.klinikum.uni-muenchen.de/Medizinische-Klinik-und-Poliklinik-II/de/index.html